CLINICAL TRIAL: NCT06466057
Title: The Efficacy of Metacognitive Therapy for Obsessive-compulsive Disorder
Brief Title: Metacognitive Therapy for Obsessive-Compulsive Disorder
Acronym: MCTOCD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Northeast Normal University (Other)
Responsible Party: Principal Investigator, Fan Jiang, Clinical Professor, Northeast Normal University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NENU2023032
Record Dates: First submitted 2024-06-13; First posted 2024-06-20 (Actual); Last update posted 2024-06-20 (Actual); Status verified 2024-06

CONDITIONS: Obsessive-Compulsive Disorder
Keywords: Obsessive-Compulsive Disorder; Metacognitive Therapy
MeSH Terms: conditions — Obsessive-Compulsive Disorder

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The outcomes assessor is a psychiatrist who was not involved in the randomization and treatment process.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Metacognitive Therapy (Experimental): Intervention using metacognitive therapy, with sessions set for 8-15 weeks of 1-2 weekly psychotherapeutic dialogue.
  Interventions: Behavioral: Metacognitive Therapy
- Control Condition (Placebo Comparator): Do not receive any additional psychotherapy in addition to conventional treatment.
  Interventions: Other: General mental health promotion

INTERVENTIONS:
Behavioral: Metacognitive Therapy — A one-on-one face-to-face dialogue format will be used to conduct psychotherapy with each participant, and the treatment protocol will be based on the treatment manual for metacognitive therapy.
  Arms: Metacognitive Therapy
Other: General mental health promotion — A general mental health mission will be conducted, not covering any metacognitive therapy related content, set for 8-15 weeks, 1 time per week
  Arms: Control Condition

SUMMARY:
The goal of this clinical trial is to learn if metacognitive therapy can be effective in a Chinese sample of obsessive compulsive disorder (OCD) . The main questions it aims to answer are:

Can metacognitive therapy significantly reduce participants' levels of obsessive-compulsive symptoms? Can metacognitive therapy significantly improve participants' metacognitive adaptations?

The researchers will compare metacognitive therapy to a control condition without psychotherapy to see if metacognitive therapy is effective in treating OCD.

Participants will:

Receive the metacognitive therapy intervention or under control conditions for 8 to 15 weeks.

Be assessed for symptoms and metacognitive beliefs at pre-intervention, post-intervention and 12 weeks post-intervention

DETAILED DESCRIPTION:
This study will be a randomised controlled clinical trial. Participants who meet the enrolment criteria will be randomised into an experimental group and a control group. Participants in the experimental group will receive 8-15 weeks of metacognitive therapy, while participants in the control group will receive the same amount of time of regular treatment without psychotherapy components.

The researchers will assess participants' obsessive-compulsive symptoms and metacognitive levels before, after, and 12 weeks after the intervention. Assessment measures will be the Yale Brown Obsessive-Compulsive Scale (Y-BOCS) and the Metacognition Questionnaire (MCQ-30).

By comparing the assessment results of the two groups of participants, conclusions will be drawn as to whether metacognitive therapy can have a positive effect on a Chinese OCD sample.

ELIGIBILITY:
Inclusion Criteria:

* two psychiatrists with the title of Deputy Chief Physician or above jointly determine that the above diagnostic criteria were met
* education level of junior high school or above, without mental retardation or audio-visual disorders
* participation in the study is voluntary, and the informed consent is signed by the patient or his/her guardian

Exclusion Criteria:

* loss of or insufficient self-awareness, the presence of hallucinations, delusions, and other psychotic symptoms
* the presence of severe depression, or self-inflicted suicidal attempts and behaviors
* the presence of a history of alcohol or drug abuse
* refusal of psychotherapy, or the ineffectiveness of those who had been involved in a full course of psychotherapy.

Ages: 12 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-06-11 (Actual); Primary Completion 2024-09-01 (Estimated); Study Completion 2024-11-01 (Estimated)

PRIMARY OUTCOMES:
Severity of participants' obsessive-compulsive symptoms | Pre-intervention to 12 weeks post-intervention
  Assessed using the Yale Brown Obsessive-Compulsive Scale (Y-BOCS) , with higher scores indicating more severe symptoms.

SECONDARY OUTCOMES:
Levels of Participants' Dysfunctional Metacognitive Beliefs | Pre-intervention to 12 weeks post-intervention
  Assessed using the Metacognition Questionnaire (MCQ-30), with higher scores being associated with more dysfunctional metacognition.

CONTACTS AND LOCATIONS:
Overall Officials: Xiaoming Liu, Ph.D, Study Director — Northeast Normal University
Locations (1):
- Northeast Normal University, Changchun, Jilin, China

IPD SHARING:
Plan to Share IPD: Yes
Data might be made available to experts in the field upon request and upon the detailed description of the reason of request.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Access to data is expected to be open by 31 January 2025 and will always be continuous.
Access Criteria: Data will be made available to experts in the field upon request and upon the detailed description of the reason of request.

REFERENCES:
- [Background] Wells A, Capobianco L, Matthews G, Nordahl HM. Editorial: Metacognitive Therapy: Science and Practice of a Paradigm. Front Psychol. 2020 Sep 18;11:576210. doi: 10.3389/fpsyg.2020.576210. eCollection 2020. No abstract available. PMID 33041948
- [Background] Fisher PL, Wells A. Metacognitive therapy for obsessive-compulsive disorder: a case series. J Behav Ther Exp Psychiatry. 2008 Jun;39(2):117-32. doi: 10.1016/j.jbtep.2006.12.001. Epub 2007 Mar 7. PMID 17418090
- See also: It contains the basic concepts of metacognitive therapy — http://evpn.library.nenu.edu.cn/piswww.frontiersin.org/journals/psychology/articles/10.3389/fpsyg.2020.576210/full
- See also: It contains a specific intervention process for metacognitive therapy — http://evpn.library.nenu.edu.cn/pislinkinghub.elsevier.com/retrieve/pii/S000579160700002X